CLINICAL TRIAL: NCT06474377
Title: A Randomized, Double-blind, Controlled Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of 24-valent Pneumococcal Conjugate Vaccine in Adults 18 Years of Age and Older
Brief Title: Clinical Trial of PCV24 in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-PCV24-1001
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Pneumococcal Infectious Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Experimental: Sinovac PCV24 formulation 1 (Experimental): 48 participants will be randomized to receive Sinovac PCV24 formulation 1. Route of administration is intramuscular injection at deltoid muscle of upper arm. Immunization schedule is 1 dose.
  Interventions: Biological: Sinovac PCV24 formulation 1
- Experimental: Sinovac PCV24 formulation 2 (Experimental): 48 participants will be randomized to receive Sinovac PCV24 formulation 2. Route of administration is intramuscular injection at deltoid muscle of upper arm. Immunization schedule is 1 dose.
  Interventions: Biological: Sinovac PCV24 formulation 2
- Active control: Pneumovax® (Active Comparator): 48 participants will be randomized to receive Pneumovax®. Route of administration is intramuscular injection at deltoid muscle of upper arm. Immunization schedule is 1 dose.
  Interventions: Biological: Pneumovax®
- Placebo: Normal saline (Placebo Comparator): 24 participants will be randomized to receive placebo. Route of administration is intramuscular injection at deltoid muscle of upper arm. Immunization schedule is 1 dose.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Sinovac PCV24 formulation 1 — One dose of Sinovac PCV24 formulation 1（0.5mL）
  Arms: Experimental: Sinovac PCV24 formulation 1
Biological: Sinovac PCV24 formulation 2 — One dose of Sinovac PCV24 formulation 2（0.5mL）
  Arms: Experimental: Sinovac PCV24 formulation 2
Biological: Pneumovax® — One dose of Pneumovax® (0.5 mL) contains 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F and 33F saccharides.
  Arms: Active control: Pneumovax®
Biological: Placebo — 0.5 mL of 0.9%NaCl solution (normal saline)
  Arms: Placebo: Normal saline

SUMMARY:
A Phase I clinical trial of 24-valent pneumococcal conjugate vaccine (PCV24) developed by Sinovac Life Science Co., Ltd will be conducted in adults aged 18 years and older. The objective of the study is to evaluate the safety and immunogenicity of Sinovac PCV24. The trial is a randomized, double-blind, controlled Phase I clinical trial.

DETAILED DESCRIPTION:
A phase I clinical trial of the study of 24-valent Pneumococcal Polysaccharide Conjugate Vaccine (PCV24) developed by Sinovac Life Science Co., Ltd (Sinovac) will be conducted in Chinese adults aged 18 years and older. The trial is a randomized, double-blind and active controlled study. The objective of this study is to evaluate the safety and immunogenicity of PCV24 manufactured by Sinovac Life Science Co., Ltd. The active control vaccine is the Pneumovax® manufactured by MSD. The placebo is 0.9%NaCl solution.

A total of at least 168 participants will be enrolled, including 84 adults aged 18-59 years and 84 elderly people aged ≥60 years. Participants will be randomized in a 2:2:2:1 ratio to receive one dose of PCV24 formulation 1, PCV24 formulation 2, Pneumovax® or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers who are aged 18 years and older, and provide legal proof of identity;
2. Participants understand and voluntarily sign the informed consent form;
3. Participants can follow all study procedures and stay in contact during the study.

Exclusion Criteria:

1. Received any pneumococcal vaccine prior to enrollment;
2. History of invasive pneumococcal diseases (IPDs) or other pneumococcal diseases caused by Streptococcus pneumoniae, as confirmed by laboratory tests;
3. History of allergy or adverse reactions to the vaccine or vaccine components, or history of allergy, such as urticaria, dyspnea, angioedema and anaphylactic shock;
4. Congenital malformations or developmental disorders, genetic defects (such as Down syndrome, thalassemia, or G6PD deficiency), severe malnutrition;
5. Have uncontrolled chronic diseases or history of severe diseases, including but not limited to cardiovascular diseases, such as hypertension uncontrolled by drugs (measurement on site: systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg) and coronary heart disease, metabolic diseases (such as uncontrolled diabetes), hematological diseases (e.g. severe anemia, hemophilia), liver and kidney diseases, digestive diseases, respiratory diseases (such as active tuberculosis), malignant tumors and major functional organ transplantation history;
6. Autoimmune diseases or immunodeficiency diseases (including but not limited to systemic lupus erythematosus, rheumatoid arthritis, autoimmune thyroid disease, asplenia, functional asplenia, HIV infection)
7. Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets level), history of obvious bleeding, hematoma or bruising after intramuscular injection or venipuncture.
8. Have/have suffered from a serious neurological disorder (epilepsy or convulsions) or mental illness or have a family history of such diseases.
9. Long-term alcohol or drug abuse.
10. Have received > 14 days of immunosuppressive or other immunomodulatory therapy (such as prednisone ≥20 mg/ day, or its equivalent) in the past 6 months, or cytotoxic therapy, or plan to receive such therapy during the study period.
11. Received immunoglobulin or other blood products within 3 months prior to enrollment, or plan to receive such treatment during the study period;
12. Received other investigational drugs or vaccines within 30 days prior to enrollment, or plan to receive such drugs or vaccines during the study;
13. Received live attenuated vaccine within 14 days prior to enrollment;
14. Received subunit or inactivated or other vaccine within 7 days prior to enrollment;
15. Acute diseases or acute onset of chronic diseases within 7 days prior to enrollment, or known or suspected active infection;
16. Women who are breastfeeding;
17. Fertile women aged 18-59 years who plan to become pregnant or cannot use effective contraception or have egg donation plans from enrollment to 3 months after the study intervention;
18. Women who are pregnant (as judged by the participant's blood pregnancy test);
19. Had fever (axillary temperature> 37.0℃) before vaccination;
20. Abnormalities in clinical laboratory indicators that exceed reference range and are clinically significant.
21. In the investigator's judgment, the participant has any other factors that make him or her unfit to participate in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions | 0-30 days after vaccination
  Incidence of adverse reactions within 30 days after vaccination

SECONDARY OUTCOMES:
Incidence of adverse reactions | 0-7 days after vaccination
  Incidence of adverse reactions within 7 days after vaccination
Incidence of serious adverse events (SAE) | 0-6 months after vaccination
  Incidence of SAE during the period of safety monitoring
Incidence of clinically significant abnormality in laboratory examination tests | 0-3 days after vaccination
  Incidence of clinically significant abnormality in blood routine, blood biochemistry and urine routine test results within 3 days after vaccination
Pneumococcal serotype-specific IgG antibody geometric mean concentration (GMC) | 30 days after vaccination
  IgG GMC 30 days after vaccination
Pneumococcal serotype-specific IgG antibody geometric mean increase (GMI) | 30 days after vaccination
  IgG GMI 30 days after vaccination
Proportion of pneumococcal serotype-specific IgG antibody concentration increase≥4 | 30 days after vaccination
  Proportion of IgG antibody concentration increase≥four folds 30 days after vaccination
Pneumococcal serotype-specific opsonophagocytic assay (OPA) geometric mean titer (GMTs) | 30 days after vaccination
  OPA GMT 30 days after vaccination
Pneumococcal serotype-specific OPA GMI | 30 days after vaccination
  OPA GMI 30 days after vaccination
Proportion of pneumococcal serotype-specific OPA antibody titer increase≥4 | 30 days after vaccination
  Proportion of OPA antibody titer increase≥four folds 30 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Kai Chu, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention (Jiangsu Provincial Academy of Preventive Medicine)
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No